CLINICAL TRIAL: NCT02339649
Title: Long-term Cognitive and Cerebral Changes in Sepsis Survivors and Their Predictors
Acronym: BonSEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Collaborators: University Hospital, Bonn (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BN005; 2011-003014-16 (EudraCT Number)
Record Dates: First submitted 2011-08-03; First posted 2015-01-15 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Severe Sepsis With Septic Shock; Severe Sepsis Without Septic Shock
Keywords: sepsis; septic shock; ICU; long-term outcome; neurocognitive; inflammatory; MRI; EEG; brain imaging; serum biomarkers; CSF
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Blood Specimen Collection; Mental Status and Dementia Tests; Spinal Puncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sepsis/septic Shock (Other): Men and women seen at the intensive care units of the Anesthesiology Department of the University Hospital Bonn aged 25-80; fulfill the criteria of sepsis and/or septic shock patients according to theThird International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3, Singer et al, 2016).
  Interventions: Neurocognitive Assessment, Clinical Scales, Questionnaires, Blood Sample, voluntary Lumbar Puncture, Resting State EEG, MRI
  Interventions: Procedure: Blood Sample; Behavioral: Neurocognitive Assessment; Other: Resting State EEG; Procedure: Lumbar Puncture; Other: MRI
- Postoperative ICU Patients (Other): Men and women seen at the intensive care units of the Anesthesiology Department of the University Hospital Bonn aged 25-80:
  * Admitted to the intensive care units of the Anesthesiological-Operative Intensive Care Unit of the University Hospital Bonn, which includes a surgical ICU, an anesthesiological ICU, and a cardio-surgical ICU
  * Duration of ICU stay must be a minimum of 24 hours.
  * Mini-Mental State Examination (MMSE) Score of 25 or above
  Interventions: Neurocognitive Assessment, Clinical Scales, Questionnaires, Blood Sample, voluntary Lumbar Puncture, Resting State EEG, MRI
  Interventions: Procedure: Blood Sample; Behavioral: Neurocognitive Assessment; Other: Resting State EEG; Procedure: Lumbar Puncture; Other: MRI
- Healthy Controls (Other): Healthy Controls will only be included in the study if they meet all of the following criteria: Written informed consent of the subject, Aged 25-80 years, Male or female.
  Interventions: Neurocognitive Assessment, Clinical Scales, Questionnaires, Blood Sample, voluntary Lumbar Puncture, Resting State EEG, MRI
  Interventions: Procedure: Blood Sample; Behavioral: Neurocognitive Assessment; Other: Resting State EEG; Procedure: Lumbar Puncture; Other: MRI

INTERVENTIONS:
Procedure: Blood Sample — Blood Sample
Behavioral: Neurocognitive Assessment — Neurocognitive Assessment
Other: Resting State EEG — 10-20 Minutes of Resting State EEG
  Other Names: Resting-State EEG
Procedure: Lumbar Puncture — Lumbar Puncture
Other: MRI — 60 Minutes MRI

SUMMARY:
The main goals of this study are to provide a cognitive, neurological, brain morphological, and serological profile of sepsis survivors in order to make long-term prognosis of recovery and estimate the need for rehabilitation measures in order to help patients reintegrate into normal daily life.

DETAILED DESCRIPTION:
Comparison of cognitive function in severe septic/septic shock ICU patients with non-septic postoperative ICU patients and actively recruited healthy controls at several time points up to 12 months after leaving the ICU.

Secondary aims:

* Profiling specific cognitive deficits in sepsis survivors over time.
* Identifying possible subclasses of long-term cognitive impairment according to facets of disease, therapy and ICU experience.
* Investigating long-term brain morphological changes, with hippocampus as region of interest (ROI).
* Determining values of Serum- and CSF-Biomarkers
* Evaluation of diagnostic and prognostic value of non-routine biomarkers for systemic- and neuroinflammation in the acute phase and in the long-term
* Investigate associations between brain morphological changes, cognitive changes, neurological status, psychiatric burden, disability level, employment status and health-related quality of life (HRQOL).
* Investigating brain-activity changes in resting state electro-encephalogram (EEG)

ELIGIBILITY:
INCLUSION CRITERIA:

sepsis/septic shock subjects will only be included in the study if they meet all of the following criteria:

* Written informed consent of the subject. or legal representative patient at the Anesthesiological-Operative Intensive Care Unit of the University Hospital Bonn, the Department of Anesthesiology, Intensive Care and Pain Therapy of the Malteser Hospital, or the Department of Anesthesiology, Intensive Care Medicine and Pain Medicine of the Gemeinschaftskrankenhaus Bonn St. Petrus Hospital. At the Anesthesiological-Operative Intensive Care Unit of the University Hospital Bonn, only, or 1) documentation of presumed will via a relative or legal representative . together with 2) Documentation of verification by a doctor independent of the study that the patient's study participation is unobjectionable. Written informed consent of patient will be obtained at the earliest time possible.
* Aged 25-80 years
* Male or female
* Admitted to the intensive care units of the Anesthesiological-Operative Intensive Care Unit of the University Hospital Bonn, from the Department of Anesthesiology, Intensive Care and Pain Therapy of the Malteser Hospital or from the Department of Anesthesiology, Intensive Care Medicine and Pain Medicine of the Gemeinschaftskrankenhaus Bonn St. Petrus Hospital.
* Duration of ICU stay must be a minimum of 24 hours. In case of transfer to intermediate care or the observation ward before the 24 hour ICU period is complete, study parameters must be allowed to be assessed.
* Fulfill the criteria of sepsis and/or septic shock patients according to theThird International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3, Singer et al, 2016).

Postoperative ICU Patients will only be included in the study if they meet all of the following criteria:

* Written informed consent of the subject.
* Aged 25-80 years
* Male or female
* Admitted to the intensive care units of the Anesthesiological-Operative Intensive Care Unit of the University Hospital Bonn, which includes a surgical ICU, an anesthesiological ICU, and a cardio-surgical ICU
* Duration of ICU stay must be a minimum of 24 hours. In case of transfer to intermediate care or the observation ward before the 24 hour ICU period is complete, study parameters must be allowed to be assessed.
* Mini-Mental Status Examination (MMSE) Score of 25 or above

Healthy Controls will only be included in the study if they meet all of the following criteria:

* Written informed consent of the subject
* Aged 25-80 years
* Male or female

EXCLUSION CRITERIA:

Subjects presenting with any of the following exclusion criteria may not be included in the study:

* Simultaneous participation in any clinical treatment study involving administration of an investigational medicinal product within 30 days prior to study beginning
* Physical or psychiatric condition which at the investigator's discretion may put the subject at risk, may confound the study results, or may interfere with the subject's participation in this study
* Prior to the start of this study existence of preexisting severe diseases and/or conduction of surgery necessarily imply life expectancy less than 12 months
* Known or suspected persistent abuse of medication, drugs or alcohol now or in the past
* Known cerebral lesions, cerebral infarction or malignomas
* Dementia or history of other central nervous system diseases
* Cranial-cerebral injury
* Known HIV-Infection
* Known liver cirrhosis with a documented Child-Pugh Score of C prior to this study
* Liver transplants
* Prior to start of this study nursing care level of 2 or 3
* Prior to start of this study residing in a nursing home

Additional Exclusion Criteria For Non-Septic Postoperative ICU Patients:

* Fulfill the criteria of sepsis and/or septic shock patients according to theThird International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3, Singer et al, 2016).
* In the case that a postoperative ICU patient fulfills the criteria for sepsis during ICU stay, he/she will be moved to the sepsis group.

Additional Exclusion Criteria For Healthy:

* Executing third-party cognitive and functional assessments of another patient-subject also included in this investigation
* History of ICU stay in the last 12 months

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Verbal Learning Memory Test Long Delayed Recall (Trial 7) | 6 months post ICU
  Verbal Learning Memory Test Long Delayed Recall (Trial 7) at 6 months post ICU admission in sepsis/septic shock patients versus non-septic postoperative patients, and comparison to actively recruited healthy controls)

SECONDARY OUTCOMES:
Verbal Learning Memory Test, German Version | For patient groups: 6 months; for Healthy Controls: Baseline
  Verbal Learning and Memory: Verbal Learning Memory Test, German Version
Verbal Learning Memory Test, German Version | For patient groups: 12 months; for Healthy Controls: 6 months
  Verbal Learning and Memory: Verbal Learning Memory Test, German Version
Wechsler Memory Scale IV Visual Recall I and II | For patient groups: 6 months; for Healthy Controls: Baseline
  Visual Memory: Wechsler Memory Scale IV Visual Recall I and II
Wechsler Memory Scale IV Visual Recall I and II | For patient groups: 12 months; for Healthy Controls: 6 months
  Visual Memory: Wechsler Memory Scale IV Visual Recall I and II
Wechsler Memory Scale Digit-Span | For patient groups: 6 months; for Healthy Controls: Baseline
  Working Memory: Wechsler Memory Scale Digit-Span
Wechsler Memory Scale Digit-Span | For patient groups: 12 months; for Healthy Controls: 6 months
  Working Memory: Wechsler Memory Scale Digit-Span
German Vocabulary Test | For patient groups: 6 months; for Healthy Controls: Baseline
  Premorbid Verbal Ability: German Vocabulary Test Mehrfachwahl Wortschatztest B (MWT-B)
German Vocabulary Test | For patient groups: 12 months; for Healthy Controls: 6 months
  Premorbid Verbal Ability: German Vocabulary Test
Symbol Digit Modalities Test | For patient groups: 6 months; for Healthy Controls: Baseline
  Cognitive Speed
Symbol Digit Modalities Test | For patient groups: 12 months; for Healthy Controls: 6 months
  Cognitive Speed
Trail Making Test A & B | For patient groups: 6 months; for Healthy Controls: Baseline
  Simple and Divided Attention
Trail Making Test A & B | For patient groups: 12 months; for Healthy Controls: 6 months
  Simple and Divided Attention
Phonetic and Lexical Verbal Fluency | For patient groups: 6 months; for Healthy Controls: Baseline
  Phonetic and Lexical Verbal Fluency
Phonetic and Lexical Verbal Fluency | For patient groups: 12 months; for Healthy Controls: 6 months
  Phonetic and Lexical Verbal Fluency
Patient Health Questionnaire Subtests Depression, Anxiety and Somatic Symptoms | For patient groups: 6 months; for Healthy Controls: Baseline
  Depression and Anxiety Inventory
Patient Health Questionnaire Subtests Depression, Anxiety and Somatic Symptoms | For patient groups: 12 months; for Healthy Controls: 6 months
  Depression and Anxiety Inventory
Post-Traumatic Stress Syndrome 10 | For patient groups: 6 months; for Healthy Controls: Baseline
  Post-Traumatic Stress Screening
Post-Traumatic Stress Syndrome 10 | For patient groups: 12 months; for Healthy Controls: 6 months
  Post-Traumatic Stress Screening
European Quality of Life 5 Dimensions-5 Levels | For patient groups: 6 months; for Healthy Controls: Baseline
  Quality of Life
European Quality of Life 5 Dimensions-5 Levels | For patient groups: 12 months; for Healthy Controls: 6 months
  Quality of Life
Functional Activities Questionnaire | For patient groups: 6 months; for Healthy Controls: Baseline
  Activities of Daily Living
Functional Activities Questionnaire | For patient groups: 12 months; for Healthy Controls: 6 months
  Activities of Daily Living
modified version of Rankin Scale Structured Interview (modified for ICU patients) | For patient groups: 6 months; for Healthy Controls: Baseline
  Function Scale
modified version of Rankin Scale Structured Interview (modified for ICU patients) | For patient groups: 12 months; for Healthy Controls: 6 months
  Function Scale
Pittsburgh Sleep Quality Index | For patient groups: 6 months; for Healthy Controls: Baseline
  Sleep Quality
Pittsburgh Sleep Quality Index | For patient groups: 12 months; for Healthy Controls: 6 months
  Sleep Quality
Mini Mental Status Examination | For patient groups: (OP Probands 1-28 d before OP, 6 months; for Healthy Controls: Baseline
  Cognitive Screening
Mini Mental Status Examination | For patient groups: 12 months; for Healthy Controls: 6 months
  Cognitive Screening
Clinical Scales at ICU | For Patients during ICU Stay (Day 0, [Day 7 if still on ICU], Day of Release)
  Therapeutic Intervention Scoring System-10, Total Score Simplified Acute Physiology Score, Sequential Organ Failure Assessment Confusion Assessment Method for the ICU
Neurological Examination | For patient groups: 6 months, 12 months; for Healthy Controls: Baseline and 6 months
  Subscales Motor ability, Walking and Standing, Behavior, Praxis/Visual or Visuospatial, Speaking and Language, Autonomic Nervous System, Tone and Muscle Exam, Coordination and Movement
resting state electroencephalogram | For patient groups: 6 months, 12 months; for Healthy Controls: Baseline and 6 months
  10-20 system electroencephalogram (64 channels with additional electro-oculogram, electromyogram, electrocardiogram). The protocol includes 5 phases, each one minute long: 1) eyes open, relaxed state, fixation of a black dot at 2 m distance, 2) word generation using letter "P" with eyes closed, 3) mental arithmetic: continuous subtraction of 7 starting from 1,000 with eyes closed, 4) eyes closed, relaxed state, no task, 5) visualization of a previously memorized geometric figure with eyes closed. Data sampled at a rate of 256 Herz using an anti-aliasing low pass filter. Power spectra will be calculated for consecutive 4-second windows and calculated for each electrode contact. Absolute spectral power will be determined for the delta (0.5-4 Herz), theta (4-8 Herz), alpha (8-13 Herz), beta (13-20 Herz) and gamma (20-40 Herz) bands, which will be averaged across all windows.
MRI (3 Tesla) of brain with hippocampus as Region of Interest | For patient groups: 6 months, 12 months; for Healthy Controls: Baseline and 6 months
  MRI (3 Tesla) of brain with hippocampus as Region of Interest. Protocol includes: three-dimensional, T1-weighted rapid gradient echo sequence, Resting State, Gradient Echo-Field-Map for Resting State, Inversion Recovery Echo Planar Imaging for Resting State, Spoiled Gradient Echo, Fluid Attenuated inversion Recovery, Susceptibility weighted imaging, Diffusion Tensor Imaging, Gradient Echo-Field-Map for Diffusion Tensor Imaging
Blood Sample | For Patient Groups 2-3 samples during ICU, 3-4 Months, 6 months, 12 Months
  All blood samples shall be drawn, stored and analyzed according to the participant information in the laboratories of the Biomarker Dementia Working Group and the Central Laboratory. Blood sampling analysis will include leukocyte count, hemoglobin, hematocrit, erythrocytes, Mean Corpuscular Hemoglobin, Meam Corpuscular Volume, mean Corpuscular Hemoglobin Concentration, Thrombocytes, Glucose, Lactate, electrolytes Sodium, Potassium, Calcium, Cholesterine, Tumor necrosis Factor-alpha, Interleukin-1 alpha, Interleukin-1 beta, Interleukin-6, C-reactive protein, Neuron Specific Enolase, Procalcitonin, S-100 Protein, as well as DNA and serum biorepository for further scientific analysis.
Lumbar Puncture (voluntary) | For Patients: (while at ICU, if clinically indicated as part of clinical routine and only if patient directly gives informed consent), 12 months; For Healthy Controls: Baseline and 6 months
  Cerebrospinal fluid (CSF) routine parameters will be analyzed by the Central Laboratory. Results will then be provided to the investigator. For determination of τ, phospho-τ, β-amyloid 1 40 and β-amyloid 1 42, 5 ml of cerebral-spinal-fluid will be analyzed at the laboratories of the German Center for Neurodegenerative Diseases (DZNE), Biomarker Dementia Working Group, Sigmund-Freud-Str. 25, 53105 Bonn

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Heneka, M.D., Principal Investigator — German Center for Neurodegenerative Diseases (DZNE); Andreas Hoeft, M.D., Study Chair — Department of Anesthesiology and Intensive Care Medicine, University Hospital Bonn; Christian Putensen, M.D., Study Chair — Research Unit Pulmonary Dysfunction and Sepsis, Department of Anesthesiology and Intensive Care Medicine, University Hospital Bonn; Thomas Klockgether, M.D., Study Chair — German Center for Neurodegenerative Diseases (DZNE)
Locations (2):
- Germany (2):
  - DZNE Center for Clinical Research, Bonn, North Rhine-Westphalia
  - Department of Anesthesiology, University Hospital Bonn, Bonn, North Rhine-Westphalia (nrw)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weberpals M, Hermes M, Hermann S, Kummer MP, Terwel D, Semmler A, Berger M, Schafers M, Heneka MT. NOS2 gene deficiency protects from sepsis-induced long-term cognitive deficits. J Neurosci. 2009 Nov 11;29(45):14177-84. doi: 10.1523/JNEUROSCI.3238-09.2009. PMID 19906966
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Semmler A, Widmann CN, Okulla T, Urbach H, Kaiser M, Widman G, Mormann F, Weide J, Fliessbach K, Hoeft A, Jessen F, Putensen C, Heneka MT. Persistent cognitive impairment, hippocampal atrophy and EEG changes in sepsis survivors. J Neurol Neurosurg Psychiatry. 2013 Jan;84(1):62-9. doi: 10.1136/jnnp-2012-302883. Epub 2012 Nov 7. PMID 23134661
- [Background] Sonneville R, Verdonk F, Rauturier C, Klein IF, Wolff M, Annane D, Chretien F, Sharshar T. Understanding brain dysfunction in sepsis. Ann Intensive Care. 2013 May 29;3(1):15. doi: 10.1186/2110-5820-3-15. PMID 23718252
- [Background] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258
- [Background] Widmann CN, Heneka MT. Long-term cerebral consequences of sepsis. Lancet Neurol. 2014 Jun;13(6):630-6. doi: 10.1016/S1474-4422(14)70017-1. PMID 24849863
- [Background] Widmann CN, Schewe JC, Heneka MT. Sepsis-associated encephalopathy versus sepsis-induced encephalopathy--authors' reply. Lancet Neurol. 2014 Oct;13(10):968-9. doi: 10.1016/S1474-4422(14)70204-2. No abstract available. PMID 25231518
- [Background] Lindlau A, Widmann CN, Putensen C, Jessen F, Semmler A, Heneka MT. Predictors of hippocampal atrophy in critically ill patients. Eur J Neurol. 2015 Feb;22(2):410-5. doi: 10.1111/ene.12443. Epub 2014 Apr 12. PMID 24724819
- See also: German Center for Neurodegenerative Disease (DZNE) — http://www.dzne.de
- See also: Department of Anesthesiology, University Hospital Bonn — http://www.kai.uni-bonn.de/